CLINICAL TRIAL: NCT00662181
Title: Follow-up on the HIGH: Low Study - the Longterm Effect of Growth Hormone
Brief Title: Follow-up on the HIGH: Low Study - the Longterm Effects of Growth Hormone
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Forskningschef Ove Andersen, Klinisk Forskningscenter, Hvidovre Hospital
Other Study IDs: H-B-2008-053; 2008-41-2145
Record Dates: First submitted 2008-04-16; First posted 2008-04-21 (Estimated); Last update posted 2008-04-21 (Estimated); Status verified 2008-04

CONDITIONS: HIV Infections; HIV-Associated Lipodystrophy Syndrome
Keywords: growth hormone; quality of life; fat redistribution; sugar metabolism; fat metabolism; cytokines
MeSH Terms: conditions — HIV Infections; HIV-Associated Lipodystrophy Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- H, NH: HIV positive patients with and without lipodystrophy

SUMMARY:
A follow-up study on the randomized, controlled, double-blind HIGH: low study. We will examine the participants from the HIGH: low study min. 6 months after finishing the HIGH: low study. We will look at the parameters: quality of life, sugar-metabolism, fat-metabolism, fat-redistribution and cytokines. The study will use the participants control visit, and the only additional examination will be the danish MOS-HIV questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years of age
* Participated in and completed the HIGH: low study
* informed consent signed

Exclusion Criteria:

* Patient stopped at Hvidovre Hospital, or didn't finish the HIGH: low study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants from the HIGH: low study
Sampling Method: Non-Probability Sample
Enrollment: 46 (Estimated)
Dates: Start 2008-05; Primary Completion 2008-10 (Estimated); Study Completion 2009-01 (Estimated)

PRIMARY OUTCOMES:
Quality of life | 6 months follow-up

SECONDARY OUTCOMES:
Metabolism | 6 months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Ove Andersen, MD, Principal Investigator — Klinisk Forskningcenter, Hvidovre Hospital
Locations (1):
- Klinisk Forskningscenter, Hvidovre Hospital, Hvidovre, Hvidovre, Denmark

REFERENCES:
- See also: The official website for Hvidovre Hospital — http://www.hvidovrehospital.dk